CLINICAL TRIAL: NCT06308822
Title: MATCH Treatment Subprotocol K1: Phase 2 Study of JNJ-42756493 (Erdafitinib) in Patients With Tumors With FGFR Amplifications
Brief Title: Testing JNJ-42756493 (Erdafitinib) as Potentially Targeting Treatment in Cancers With FGFR Amplifications (MATCH-Subprotocol K1)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01151; NCI-2024-01151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-K1 (Other: ECOG-ACRIN Cancer Research Group); EAY131-K1 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-03-09; First posted 2024-03-13 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; erdafitinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (erdafitinib) (Experimental): Patients receive erdafitinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout study. Patients may also undergo blood sample collection and tumor biopsy throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Erdafitinib; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II MATCH treatment trial tests how well JNJ-42756493 (erdafitinib) works in treating patients with tumors that have more copies of the FGFR gene than is normal (amplification). Erdafitinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal FGFR protein that signals cancer cells to multiply.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive erdafitinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout study. Patients may also undergo blood sample collection and tumor biopsy throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol.
* Patients must fulfill all eligibility criteria outlined in MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7).
* Patients must have FGFR Amplification as determined via the MATCH Master Protocol.
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block).
* Patients must not have known hypersensitivity to JNJ-42756493 (erdafitinib) or compounds of similar chemical or biologic composition.
* Patients with current evidence of corneal or retinal disorder/keratopathy are excluded.
* Patients must not be currently using medications that can elevate serum phosphorous and/or calcium levels.

  * Medications that increase serum calcium should be avoided. Over the counter calcium supplements, antacids that contain calcium (Tums) and vitamin D supplements (cholecalciferol and ergocalciferol) should be avoided. Prescription medications including lithium, hydrochlorothiazide and chlorthalidone must be used with caution.
  * Medications that increase serum phosphate should be avoided. Over the counter laxatives that contain phosphate such as Fleets oral or Fleets enema and Miralax should be avoided.
* Patients with a history of hyperphosphatemia will be excluded.
* Patients may not have received strong inhibitors or potent inducers of CYP3A within 2 weeks before the first dose of study treatment. Patients with inability to discontinue treatment with a strong CYP3A4 and/or CYP2C9 inhibitor or inducer prior to start of treatment are excluded.
* Patients who have previously received treatment with a FGFR-targeted inhibitor are excluded. Such inhibitors include AZD4547, BGJ398, BAY1163877 and LY2874455). Prior non-selective FGFR inhibitor treatment (e.g. Pazopanib, dovitinib, ponatinib, brivanib, lucitanib, lenvatinib) are allowed.
* Patients must not have any history of or current evidence of renal or endocrine alterations of calcium/phosphate homeostasis, or history of or current evidence of extensive tissue calcification (by evaluation of the clinician), including but not limited to, the soft tissue, kidneys, intestine, myocardium and lung with the exception of calcified lymph nodes and asymptomatic vascular calcification per investigators' judgment.
* Patients with transitional cell carcinoma of the bladder and /or urothelial tract are not eligible. These patients are encouraged to enroll in the ongoing disease-specific studies.
* Patients with impaired renal function (glomerular filtration rate [GFR] < 60 mL/min) are excluded. GFR should be assessed by direct measurement (i.e., creatinine clearance or ethyldediaminetetraacetate) or, if not available, by calculation from serum/plasma creatinine (Cockcroft-Gault formula).
* Patients with persistent phosphate level > upper limit of normal (ULN) during screening (within 14 days of treatment and prior to cycle 1 day 1) and despite medical management are excluded.
* Patients with a history of or current uncontrolled cardiovascular disease as stated below are excluded:

  * Unstable angina, myocardial infarction, or known congestive heart failure class II-IV within the preceding 12 months; cerebrovascular accident or transient ischemic attack within the preceding 3 months, pulmonary embolism within the preceding 2 months.
  * Any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, cardiac arrest, Mobitz II second degree heart block or third degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy.
* Patients with impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions are excluded.
* Female subjects (of child-bearing potential and sexually active) must use medically acceptable methods of birth control (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of the study, and for 4 months after the last intake of study drug. Male subjects (with a partner of child-bearing potential) must use a condom with spermicide when sexually active and must not donate sperm from the first dose of study drug until 5 months after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alain C Mita, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on June 20, 2018. Thirty-five patients were enrolled between August 20, 2018, and April 30, 2019.
Pre-assignment Details: The FGFR amplification status was determined by assay performed in a NCI-MATCH approved laboratory for all patients in this arm. Mutation status was confirmed by central MATCH assay for 18 patients.
Groups:
- Treatment (Erdafitinib): Patients receive erdafitinib 8 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout study. Patients may also undergo blood sample collection and tumor biopsy throughout the trial.
Period: Overall Study
Arm/Group | Treatment (Erdafitinib)
Started | 35
Eligible | 34
Started Protocol Therapy | 34
Eligible and Treated | 33
Mutation Status Confirmed | 18
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis population) | 18
Completed (Treatment continued until disease progression or intolerability) | 0
Not Completed | 35
Not completed — Mutation Status Not Confirmed | 17
Not completed — Adverse Event | 1
Not completed — Death | 5
Not completed — Disease progression | 8
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable (ie, eligible, treated and PIK3CA mutation status confirmed) patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 18
percentage of participants | 0 [0 to 15.3]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 18
percentage of participants | 13.8 [3.3 to 31.6]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Erdafitinib)
Number analyzed (Participants) | 18
months | 1.7 [1.1 to 1.8]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-three patients were included in the toxicity analysis (excluding one never treated and one without toxicity data collected).
Arm/Group | Treatment (Erdafitinib)
All-Cause Mortality (participants affected / at risk) | 32/35
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erdafitinib) (N=33)
Anemia (Blood and lymphatic system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erdafitinib) (N=33)
Anemia (Blood and lymphatic system disorders) | 4
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 15
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 2
Investigations - Other, specify (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 6
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT06308822/Prot_001.pdf